CLINICAL TRIAL: NCT06338332
Title: Obstructive Colon Cancer, a Bridge to Surgery in Right Sided Obstructive Colon Cancer
Acronym: OCCBRIGHT
Status: Recruiting | Type: Observational
Sponsor: Amphia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AW23.050, W19.249
Record Dates: First submitted 2024-03-07; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-02

CONDITIONS: Colonic Neoplasms Malignant
Keywords: Right-sided; Bridge-to-surgery; Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nasogastric tube: Patients with right sided obstructive colon cancer will receive non-surgical decompression with a nasogastric probe. Prior to the definitive oncological resection, patients undergo preoperative optimisation which involves the engagement of a dietician and physiotherapist. Patients eligible for elective resection will have their resection 7-10 days after initial decompression.
- Ileostomy: Patients with right sided obstructive colon cancer will receive a ileostomy. Prior to the definitive oncological resection, patients undergo preoperative optimisation which involves the engagement of a dietician and physiotherapist. Patients eligible for elective resection will be operated at least 7 days after initial decompression and no later than 4 weeks after initial presentation.
- Right-sided stent: Patients with right sided obstructive colon cancer will receive a right-sided stent. Prior to the definitive oncological resection, patients undergo preoperative optimisation which involves the engagement of a dietician and physiotherapist. Patients eligible for elective resection will be operated at least 7 days after initial decompression and no later than 4 weeks after initial presentation.

SUMMARY:
Rationale: Approximately 13% (range 10-28%) of all colorectal cancer patients (CRC) present with an acute obstruction. Postoperative mortality after an emergency resection is known for its high risk of morbidity and mortality. Different options can be considered in the management of obstructing right sided CRC: 1) primary resection, simultaneous treatment of obstruction and tumour resection, or 2) staged treatment of the obstruction with secondary resection of the tumour. Currently, in the Netherlands, an emergency resection has been judged to be inferior to postponing surgery. Patients who present with right sided obstructive colon cancer at one of the participating hospitals are subjected to a bridge to surgery (BTS) protocol.

Objective: The primary objective of this study is to determine the feasibility of BTS protocols in right sided obstructive colon cancer and reduce mortality- and morbidity (stoma rates, major- and minor complications) rates in potentially curable patients presenting with acute obstructing colon cancer.

Study design: This is a multicentre, prospective registration study Study population: All patients presenting with high clinical suspicion or histologically proven right sided colon cancer and signs of obstruction of the large bowel.

Intervention: Prospective registration of the implementation of bridge to surgery protocols in patients with (acute) malignant right sided obstruction of the colon, without suspicion of perforation (tumour perforation or blow out) in order to optimize patients preoperatively. The BTS approach encompasses the utilization of either ileostomy creation, stent placement or nasogastric tube for decompression, which is subsequently followed by definitive surgical treatment at a later stage. BTS also involves pre-optimization, prior to the surgical procedure, with the following approach: optimizing the nutritional health status improving the physical health status of the patient.

Main study parameters/endpoints: The primary endpoint is complication-free survival (CFS) at 90 days after hospitalization. Complication is defined here as mortality and/or development of a major complication (Clavien-Dindo classification ≥3). With a total follow up of three years. Secondary endpoints: overall mortality, morbidity (stoma rates, minor complications), in hospital stay, oncologic quality of resection and other occurring adverse events.

DETAILED DESCRIPTION:
Approximately 13% (range 8-28%) presents with acute obstructing colorectal cancer (CRC). It's known that patients with acute obstructing CRC have increased mortality and morbidity compared to patients without acute obstructing CRC. Postoperative mortality ranges from 12 to 30%, which can raise to 41% in elderly patients with two or more additional risk factors. Morbidity rates until 78% are described in older patients undergoing emergency resection for obstructing CRC.

Different treatment options have been evaluated over the years. The two main options are; 1) emergency resection, simultaneous treatment of obstruction and tumour resection, 2) staged treatment of the obstruction with secondary resection of the tumour. Postoperative mortality after an emergency resection is known for its high risk of morbidity and mortality. From the Dutch audits it is know that the risk is high, not only for left sided obstruction, but also for right sided obstruction. Until recently, an acute emergency resection was the standard treatment for patients presenting with a small bowl ileus caused by a right sided colon cancer. However, more evidence has emerged that postponing surgery with a bridge tot surgery protocol can be beneficial to the patients. The bridge to surgery approach encompasses the utilization of either ileostomy creation or stent placement for colonic decompression, which is subsequently followed by definitive surgical treatment at a later stage. Alternatively, BTS may involve the introduction of a pause, also known as preoptimization, prior to the surgical procedure. The three main options for staged surgery all have its own up- and downsides. All forms of staged treatment appears to lead to fewer morbidity and mortality.

Emergency surgery Emergency resection is associated with a high risk of mortality and morbidity. Besides that, stoma creations after emergency surgery are higher than in patients treated electively. In case of a Hartmann's procedure, (resection of a left-sided tumour and creation of a colostomy) second surgical procedure is needed to restore continuity. Continuity restore has a mean mortality of 1% (range 0-7.4%) and morbidity of 16% (range 3-50%). Alternatively, emergency resection with primary anastomosis, which has the advantage to be a definite procedure, is performed. However, this treatment can be complicated with anastomotic leakage (AL). Anastomotic leakage is higher in patients treated for obstructing CRC in comparison with staged or electively treatment. Besides that, mortality rates after anastomotic leakage after colorectal surgery varies between 5-19%. Therefore, this intervention does not align with existing treatment strategies.

Bridge to surgery Stoma creation for colonic decompression followed by definite surgical treatment in a later stadium for patients with obstructing right sided CRC is an alternative. Postoperative mortality between patients treated with emergency resection, stent or stoma followed by resection showed no differences. However, high mortality rates in elderly patients (30%) after acute resection, stress the need for alternative strategies. For right-sided colon cancer, postoperative complications for patients treated with decompressing stoma before resection are lower in comparison with acute resection. However, the creation of an ileostomy leads to a longer hospital stay. Secondly, stenting as a bridge to surgery (BTS) creates time before definite surgical treatment. However, the use of stents as a bridge to surgery has controversial results. Stents as a BTS is associated with complications like perforation, stent migration, higher recurrence rate and re-obstruction. Furthermore, three prospective trials are closed prematurely because of high morbidity rates or a high number of technical failure of the self-expandable metallic stent (SEMS) However, several studies and one meta-analysis show promising short-term outcomes for the use of stents as BTS. Besides that, promising long-term outcomes, such as oncological safety, after stents as BTS are shown. Finally, transtumoral intubation for decompression of the colon, before initial can be considered to prevent stoma creation. Thirdly, a bridge to surgery may involve the introduction of a pause, also known as preoptimization, prior the surgical procedure. This previously presented as PRE-OCC, this approach appears feasible and safe. Deteriorating physical condition caused by poor intake, vomiting, changes in electrolyte status and weight loss often results in a decreased nutritional status. Nutritional status and thereby the patients preoperative health status seems to influence the mortality risk for patients with (obstructing) colorectal cancer. Creating a pause, before surgery provides a chance to optimise the patients' medical condition, perform a complete pre-operative screening of the patient's health status and examine possible concomitant illnesses. Besides nutritional status, also the functional capacity of the patient seems to be an important factor in postoperative mortality and morbidity. Studies, in elective colorectal surgery, show promising results after improving the functional capacity of patients (prehabilitation) on the recovery after colorectal surgery. However, this third option of bridge to surgery also has some disadvantages. Preoptimization leads to an prolonged duration of stay prior to surgery in a semi acute setting, with a central venous line and potentially insufficient decompression.

This study aims to determine whether implementation of bridge to surgery protocols is feasible and reduces mortality- and morbidity (stoma rates, major- and minor complications) rates in potentially curable patients presenting with acute obstructing CRC. By prospectively collecting the data, the feasibility of the protocols will be reported and the decrease in mortality and morbidity rates can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is 18 years or older
* Patients presenting with symptoms of obstruction (including cecum, ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid colon) caused by (high suspicion or histologically proven) colonic cancer.
* Patient presenting with symptoms of partial obstruction (abdominal pain, nausea, vomiting, diarrhoea) confirmed by the presence of a dilated colon or ileum with a computed tomography (CT-scan).
* Treatment with curative intent.

Exclusion Criteria:

* Obstruction of the colon pathologically caused by benign disease.
* Obstruction of the colon caused by an extra-colonic malignancy.
* Suspicion of emergency complications caused by peritonitis due to perforation (tumour or blow out) or sepsis.
* Patients with advanced disease who will undergo a palliative trajectory.
* Rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with high clinical suspicion of malignant obstruction of the right sided large bowel.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Complication-free survival | 90 days after hospitalization
  The primary endpoint is complication-free survival (CFS) at 90 days after hospitalization. Complication is defined here as mortality and/or development of a major complication (Clavien-Dindo classification ≥3).

SECONDARY OUTCOMES:
Complications overall | 90 days after hospitalization
  All complications (following Clavien-Dindo classification) within 90 days after hospitalisation
Type of surgical intervention | Day of surgery
  Type of surgical intervention
Time till surgery | Days from admission untill day of surgery (up to 100 days)
  Days from admission untill day of surgery
Resection | Day of the surgery
  Creation of primary anastomosis or stoma creation
TNM | Day of the surgery
  Cancer stage (clinical and pathological) according to the tumour node metastasis (TNM) classification of the American Joint Committee
Hospital stay | Days between surgery and moment of discharge (up to 100 days)
  Total hospital stay (in total, after resection or reoperation) (days)
One year stoma rate | One year postoperative
  One year stoma rate, patients with a stoma after one year
One year survival rates | One years postoperative
  One year survival rates
Disease free survival rates one year | One years postoperative
  Rate of patients with disease free survical one year postoperative based on radiological assessment
Disease free survival rates three years | Three years postoperative
  Rate of patients with disease free survical three year postoperative based on radiological assessment
Three year survival rates | Three years postoperative
  Three year survival rates
Tumour type (obstructing, not obstructing), | At time of diagnosis
  Was there an obstructive tumor?
Metastasis preoperative | At time of diagnosis
  Presence of metastases at the time of diagnosis
Pre-operative diagnostics | At time of diagnosis
  Endoscopy, CT-scan, ultrasound and/or MRI
Type of bridge-to-surgery | At time of diagnosis
  Ileostomy, stent or nasogastric tube for decompression
Nutrition (TPN/extra nutrition) | During hospital stay (up to 100 days)
  Did the patient received additional nutrition?
Consultation of other specialist | During hospital stay (up to 100 days)
  Consultation of other specialist during hospital stay

OTHER OUTCOMES:
Gender | At time of diagnosis
  male/female
Age at surgery | At time of diagnosis
  Age at surgery (years, min 18years-max 120 years)
ASA | At time of diagnosis
  American Society of Anaesthesiologists (ASA) score (I-V)
Bodyweight | At time of diagnosis
  Bodyweight at hospital presentation (kilograms, min 30 - max 150)
Height | At time of diagnosis
  Height (centimeters, min 120cm - max 230cm)
Concomitant and previous therapy | At time of diagnosis
  Concomitant and previous therapy for this tumour (chemotherapy/radiation)
C-reactive protein | During hospital stay (up to 1 week postoperative)
  C-reactive protein (CRP, mg/L) (0-500, higher score is worse)
Haemoglobin | During hospital stay (up to 1 week postoperative)
  Haemoglobin (Hb, g/dL) (1-12, lower score is worse)
Laboratory values | During hospital stay (up to 1 week postoperative)
  Hematocrit (H, %) (0-100, the normal hematocrit for men is 40 to 54%; for women it is 36 to 48%)
Leukocytes | During hospital stay (up to 1 week postoperative)
  Leukocytes (× 10^9/L), the normal range is 4.5 to 11.0 × 109/L
Prothrombin time | During hospital stay (up to 1 week postoperative)
  Prothrombin time (PTT, seconds), normal range is 11 to 13.5 seconds
Sodium | During hospital stay (up to 1 week postoperative)
  Sodium (mEq/L), normal range 135 to 145 milliequivalents per liter (mEq/L)
Potassium | During hospital stay (up to 1 week postoperative)
  Potassium (mmol/L), normal range 3.6 to 5.2 millimoles per liter
Glomerular filtration rate | During hospital stay (up to 1 week postoperative)
  Glomerular filtration rate (GFR, mL/min/1.73 m2), normal value >90
Albumin | During hospital stay (up to 1 week postoperative)
  Albumin (g/dL), normal range 3.5 to 5.5 grams per deciliter
Bilirubin | During hospital stay (up to 1 week postoperative)
  Bilirubin (µmol/L), normal value less than 5.1 µmol/L
ASAT | During hospital stay (up to 1 week postoperative)
  Alanine- Amino-Transferase (ASAT, U/L), normal range 8 to 33 U/L
ALAT | During hospital stay (up to 1 week postoperative)
  Aspartate-Amino -transferase (ALAT, U/L), normal range 4 to 36 U/L
LDH | During hospital stay (up to 1 week postoperative)
  Lactic acid dehydrogenase (LDH,U/L), normal range 140 to 280 U/L
ALP | During hospital stay (up to 1 week postoperative)
  Alkaline phosphatase (ALP, IU/L), normal range 44 to 147
Gamma-GT | During hospital stay (up to 1 week postoperative)
  Gamma-GT (U/L), normal range 0 to 30 IU/L
Creatinkinase | During hospital stay (up to 1 week postoperative)
  Creatinkinase (U/L), norman range 22 to 198
Phosphate | During hospital stay (up to 1 week postoperative)
  Phosphate (mg/dL), normal range 2.5 to 4.5
Lactate | During hospital stay (up to 1 week postoperative)
  Lactate (mg/dL), normal value <1.0

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Schreinemakers, MD, PhD, Principal Investigator — Amphia Hospital Breda, The Netherlands
Locations (1):
- Amphia Hospital, Breda, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boeding JRE, Cuperus IE, Rijken AM, Crolla RMPH, Verhoef C, Gobardhan PD, Schreinemakers JMJ. Postponing surgery to optimise patients with acute right-sided obstructing colon cancer - A pilot study. Eur J Surg Oncol. 2023 Sep;49(9):106906. doi: 10.1016/j.ejso.2023.04.005. Epub 2023 Apr 9. PMID 37061403
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] van Rooijen SJ, Molenaar CJL, Schep G, van Lieshout RHMA, Beijer S, Dubbers R, Rademakers N, Papen-Botterhuis NE, van Kempen S, Carli F, Roumen RMH, Slooter GD. Making Patients Fit for Surgery: Introducing a Four Pillar Multimodal Prehabilitation Program in Colorectal Cancer. Am J Phys Med Rehabil. 2019 Oct;98(10):888-896. doi: 10.1097/PHM.0000000000001221. PMID 31090551
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Nishiyama VKG, Albertini SM, Moraes CMZG, Godoy MF, Netinho JG. MALNUTRITION AND CLINICAL OUTCOMES IN SURGICAL PATIENTS WITH COLORECTAL DISEASE. Arq Gastroenterol. 2018 Oct-Dec;55(4):397-402. doi: 10.1590/S0004-2803.201800000-85. PMID 30785525
- [Background] Barao K, Abe Vicente Cavagnari M, Silva Fucuta P, Manoukian Forones N. Association Between Nutrition Status and Survival in Elderly Patients With Colorectal Cancer. Nutr Clin Pract. 2017 Oct;32(5):658-663. doi: 10.1177/0884533617706894. Epub 2017 May 23. PMID 28535359
- [Background] Schwegler I, von Holzen A, Gutzwiller JP, Schlumpf R, Muhlebach S, Stanga Z. Nutritional risk is a clinical predictor of postoperative mortality and morbidity in surgery for colorectal cancer. Br J Surg. 2010 Jan;97(1):92-7. doi: 10.1002/bjs.6805. PMID 20013933
- [Background] Li CY, Guo SB, Wang NF. Decompression of acute left-sided malignant colorectal obstruction: comparing transanal drainage tube with metallic stent. J Clin Gastroenterol. 2014 May-Jun;48(5):e37-42. doi: 10.1097/MCG.0b013e31829f30ca. PMID 24162168
- [Background] Shigeta K, Baba H, Yamafuji K, Kaneda H, Katsura H, Kubochi K. Outcomes for patients with obstructing colorectal cancers treated with one-stage surgery using transanal drainage tubes. J Gastrointest Surg. 2014 Aug;18(8):1507-13. doi: 10.1007/s11605-014-2541-1. Epub 2014 May 29. PMID 24871080
- [Background] Amelung FJ, Borstlap WAA, Consten ECJ, Veld JV, van Halsema EE, Bemelman WA, Siersema PD, Ter Borg F, van Hooft JE, Tanis PJ; Dutch Snapshot Research Group. Propensity score-matched analysis of oncological outcome between stent as bridge to surgery and emergency resection in patients with malignant left-sided colonic obstruction. Br J Surg. 2019 Jul;106(8):1075-1086. doi: 10.1002/bjs.11172. Epub 2019 May 10. PMID 31074507
- [Background] van den Berg MW, Sloothaak DA, Dijkgraaf MG, van der Zaag ES, Bemelman WA, Tanis PJ, Bosker RJ, Fockens P, ter Borg F, van Hooft JE. Bridge-to-surgery stent placement versus emergency surgery for acute malignant colonic obstruction. Br J Surg. 2014 Jun;101(7):867-73. doi: 10.1002/bjs.9521. Epub 2014 Apr 16. PMID 24740753
- [Background] Tan CJ, Dasari BV, Gardiner K. Systematic review and meta-analysis of randomized clinical trials of self-expanding metallic stents as a bridge to surgery versus emergency surgery for malignant left-sided large bowel obstruction. Br J Surg. 2012 Apr;99(4):469-76. doi: 10.1002/bjs.8689. Epub 2012 Jan 19. PMID 22261931
- [Background] Zhang Y, Shi J, Shi B, Song CY, Xie WF, Chen YX. Self-expanding metallic stent as a bridge to surgery versus emergency surgery for obstructive colorectal cancer: a meta-analysis. Surg Endosc. 2012 Jan;26(1):110-9. doi: 10.1007/s00464-011-1835-6. Epub 2011 Jul 26. PMID 21789642
- [Background] Alcantara M, Serra-Aracil X, Falco J, Mora L, Bombardo J, Navarro S. Prospective, controlled, randomized study of intraoperative colonic lavage versus stent placement in obstructive left-sided colonic cancer. World J Surg. 2011 Aug;35(8):1904-10. doi: 10.1007/s00268-011-1139-y. PMID 21559998
- [Background] van Hooft JE, Fockens P, Marinelli AW, Bossuyt PM, Bemelman WA; Dutch Stent-In study group. Premature closure of the Dutch Stent-in I study. Lancet. 2006 Nov 4;368(9547):1573-4. doi: 10.1016/S0140-6736(06)69660-8. No abstract available. PMID 17084754
- [Background] Sloothaak DA, van den Berg MW, Dijkgraaf MG, Fockens P, Tanis PJ, van Hooft JE, Bemelman WA; collaborative Dutch Stent-In study group. Oncological outcome of malignant colonic obstruction in the Dutch Stent-In 2 trial. Br J Surg. 2014 Dec;101(13):1751-7. doi: 10.1002/bjs.9645. Epub 2014 Oct 9. PMID 25298250
- [Background] van Hooft JE, Bemelman WA, Oldenburg B, Marinelli AW, Lutke Holzik MF, Grubben MJ, Sprangers MA, Dijkgraaf MG, Fockens P; collaborative Dutch Stent-In study group. Colonic stenting versus emergency surgery for acute left-sided malignant colonic obstruction: a multicentre randomised trial. Lancet Oncol. 2011 Apr;12(4):344-52. doi: 10.1016/S1470-2045(11)70035-3. PMID 21398178
- [Background] Pirlet IA, Slim K, Kwiatkowski F, Michot F, Millat BL. Emergency preoperative stenting versus surgery for acute left-sided malignant colonic obstruction: a multicenter randomized controlled trial. Surg Endosc. 2011 Jun;25(6):1814-21. doi: 10.1007/s00464-010-1471-6. Epub 2010 Dec 18. PMID 21170659
- [Background] Frago R, Biondo S, Millan M, Kreisler E, Golda T, Fraccalvieri D, Miguel B, Jaurrieta E. Differences between proximal and distal obstructing colonic cancer after curative surgery. Colorectal Dis. 2011 Jun;13(6):e116-22. doi: 10.1111/j.1463-1318.2010.02549.x. PMID 21564463
- [Background] Kube R, Mroczkowski P, Granowski D, Benedix F, Sahm M, Schmidt U, Gastinger I, Lippert H; Study group Qualitatssicherung Kolon/Rektum-Karzinome (Primartumor) (Quality assurance in primary colorectal carcinoma). Anastomotic leakage after colon cancer surgery: a predictor of significant morbidity and hospital mortality, and diminished tumour-free survival. Eur J Surg Oncol. 2010 Feb;36(2):120-4. doi: 10.1016/j.ejso.2009.08.011. Epub 2009 Sep 22. PMID 19775850
- [Background] Gessler B, Eriksson O, Angenete E. Diagnosis, treatment, and consequences of anastomotic leakage in colorectal surgery. Int J Colorectal Dis. 2017 Apr;32(4):549-556. doi: 10.1007/s00384-016-2744-x. Epub 2017 Jan 9. PMID 28070659
- [Background] Ramphal W, Boeding JRE, Gobardhan PD, Rutten HJT, de Winter LJMB, Crolla RMPH, Schreinemakers JMJ. Oncologic outcome and recurrence rate following anastomotic leakage after curative resection for colorectal cancer. Surg Oncol. 2018 Dec;27(4):730-736. doi: 10.1016/j.suronc.2018.10.003. Epub 2018 Oct 10. PMID 30449500
- [Background] van de Wall BJ, Draaisma WA, Schouten ES, Broeders IA, Consten EC. Conventional and laparoscopic reversal of the Hartmann procedure: a review of literature. J Gastrointest Surg. 2010 Apr;14(4):743-52. doi: 10.1007/s11605-009-1084-3. PMID 19936852
- [Background] Pisano M, Zorcolo L, Merli C, Cimbanassi S, Poiasina E, Ceresoli M, Agresta F, Allievi N, Bellanova G, Coccolini F, Coy C, Fugazzola P, Martinez CA, Montori G, Paolillo C, Penachim TJ, Pereira B, Reis T, Restivo A, Rezende-Neto J, Sartelli M, Valentino M, Abu-Zidan FM, Ashkenazi I, Bala M, Chiara O, De' Angelis N, Deidda S, De Simone B, Di Saverio S, Finotti E, Kenji I, Moore E, Wexner S, Biffl W, Coimbra R, Guttadauro A, Leppaniemi A, Maier R, Magnone S, Mefire AC, Peitzmann A, Sakakushev B, Sugrue M, Viale P, Weber D, Kashuk J, Fraga GP, Kluger I, Catena F, Ansaloni L. 2017 WSES guidelines on colon and rectal cancer emergencies: obstruction and perforation. World J Emerg Surg. 2018 Aug 13;13:36. doi: 10.1186/s13017-018-0192-3. eCollection 2018. PMID 30123315
- [Background] Amelung FJ, Consten ECJ, Siersema PD, Tanis PJ. A Population-Based Analysis of Three Treatment Modalities for Malignant Obstruction of the Proximal Colon: Acute Resection Versus Stent or Stoma as a Bridge to Surgery. Ann Surg Oncol. 2016 Oct;23(11):3660-3668. doi: 10.1245/s10434-016-5247-7. Epub 2016 May 24. PMID 27221360
- [Background] Tan KK, Sim R. Surgery for obstructed colorectal malignancy in an Asian population: predictors of morbidity and comparison between left- and right-sided cancers. J Gastrointest Surg. 2010 Feb;14(2):295-302. doi: 10.1007/s11605-009-1074-5. Epub 2009 Nov 6. PMID 19894082
- [Background] Kolfschoten NE, Wouters MW, Gooiker GA, Eddes EH, Kievit J, Tollenaar RA, Marang-van de Mheen PJ; Dutch Surgical Colorectal Audit group. Nonelective colon cancer resections in elderly patients: results from the dutch surgical colorectal audit. Dig Surg. 2012;29(5):412-9. doi: 10.1159/000345614. Epub 2012 Dec 13. PMID 23235489
- [Background] Tanis PJ, Paulino Pereira NR, van Hooft JE, Consten EC, Bemelman WA; Dutch Surgical Colorectal Audit. Resection of Obstructive Left-Sided Colon Cancer at a National Level: A Prospective Analysis of Short-Term Outcomes in 1,816 Patients. Dig Surg. 2015;32(5):317-24. doi: 10.1159/000433561. Epub 2015 Jul 4. PMID 26159388
- [Background] Aslar AK, Ozdemir S, Mahmoudi H, Kuzu MA. Analysis of 230 cases of emergent surgery for obstructing colon cancer--lessons learned. J Gastrointest Surg. 2011 Jan;15(1):110-9. doi: 10.1007/s11605-010-1360-2. Epub 2010 Oct 26. PMID 20976568
- [Background] Ho KS, Quah HM, Lim JF, Tang CL, Eu KW. Endoscopic stenting and elective surgery versus emergency surgery for left-sided malignant colonic obstruction: a prospective randomized trial. Int J Colorectal Dis. 2012 Mar;27(3):355-62. doi: 10.1007/s00384-011-1331-4. Epub 2011 Oct 28. PMID 22033810
- [Background] Panis Y, Maggiori L, Caranhac G, Bretagnol F, Vicaut E. Mortality after colorectal cancer surgery: a French survey of more than 84,000 patients. Ann Surg. 2011 Nov;254(5):738-43; discussion 743-4. doi: 10.1097/SLA.0b013e31823604ac. PMID 21997816
- [Background] Bakker IS, Snijders HS, Grossmann I, Karsten TM, Havenga K, Wiggers T. High mortality rates after nonelective colon cancer resection: results of a national audit. Colorectal Dis. 2016 Jun;18(6):612-21. doi: 10.1111/codi.13262. PMID 26749028
- [Background] Boeding JRE, Ramphal W, Crolla RMPH, Boonman-de Winter LJM, Gobardhan PD, Schreinemakers JMJ. Ileus caused by obstructing colorectal cancer-impact on long-term survival. Int J Colorectal Dis. 2018 Oct;33(10):1393-1400. doi: 10.1007/s00384-018-3132-5. Epub 2018 Jul 25. PMID 30046958
- [Background] Jullumstro E, Wibe A, Lydersen S, Edna TH. Colon cancer incidence, presentation, treatment and outcomes over 25 years. Colorectal Dis. 2011 May;13(5):512-8. doi: 10.1111/j.1463-1318.2010.02191.x. PMID 20128833
- [Background] Van Leersum NJ, Snijders HS, Henneman D, Kolfschoten NE, Gooiker GA, ten Berge MG, Eddes EH, Wouters MW, Tollenaar RA; Dutch Surgical Colorectal Cancer Audit Group; Bemelman WA, van Dam RM, Elferink MA, Karsten TM, van Krieken JH, Lemmens VE, Rutten HJ, Manusama ER, van de Velde CJ, Meijerink WJ, Wiggers T, van der Harst E, Dekker JW, Boerma D. The Dutch surgical colorectal audit. Eur J Surg Oncol. 2013 Oct;39(10):1063-70. doi: 10.1016/j.ejso.2013.05.008. Epub 2013 Jul 18. PMID 23871573